CLINICAL TRIAL: NCT06380205
Title: A Phase 1, Open-Label Study to Evaluate the Drug Interaction Between Povorcitinib and the Oral Contraceptive Levonorgestrel/Ethinyl Estradiol in Healthy Adult Females
Brief Title: A Study to Evaluate the Drug Interaction Between Povorcitinib and the Oral Contraceptive Levonorgestrel/Ethinyl Estradiol in Healthy Adult Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB54707-111
Record Dates: First submitted 2024-04-03; First posted 2024-04-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Healthy Participants
Keywords: INCB054707
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Povorcitinib + levonorgestrel (LNG)/ethinyl estradiol (EE) (Experimental): Povorcitinib and LNG/EE will be administered at the protocol defined doses.
  Interventions: Drug: Povorcitinib; Drug: Levonorgestrel/Ethinyl estradiol

INTERVENTIONS:
Drug: Povorcitinib — Povorcitinib will be administered at protocol defined dose.
  Other Names: INCB054707
Drug: Levonorgestrel/Ethinyl estradiol — Levonorgestrel/Ethinyl estradiol will be administered at protocol defined dose.

SUMMARY:
The purpose of this study is to evaluate the drug interaction between povorcitinib and the oral contraceptive levonorgestrel/ethinyl estradiol in healthy adult females.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Females aged 18 to 60 years, inclusive, at the time of signing the ICF.
* Body mass index between 18.0 and 30.5 kg/m2, inclusive.
* No clinically significant findings in screening evaluations (eg, clinical, laboratory, and ECG evaluations).
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months before screening.
* Presence or history of a malabsorption syndrome (eg, Crohn's disease or chronic pancreatitis) that could affect drug absorption.
* Current or recent (within 3 months before screening) clinically significant gastrointestinal disease (eg, gallbladder disease) or surgery (including cholecystectomy; excluding appendectomy) that could affect the absorption of study treatment.
* History of cardiovascular, cerebrovascular, peripheral vascular, or thrombotic disease (eg, deep vein thrombosis), pulmonary embolism, or uncontrolled hypertension (ie, blood pressure > 140/90 mmHg at screening, confirmed by repeat testing).
* Positive test for HBV, HCV, or HIV. Participants whose results are compatible with prior immunization for or immunity due to infection with HBV may be included at the discretion of the investigator.
* History of tobacco- or nicotine-containing product-use within 1 month before screening.
* Pregnant, breastfeeding, or planning to conceive during the study.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Levonorgestrel (LNG) concentration in plasma | Up to Day 21
  LNG concentration in plasma.
Ethinyl estradiol (EE) concentration in plasma | Up to Day 21
  EE concentration in plasma.

SECONDARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 32
  Defined as any adverse event, either reported for the first time or the worsening of a pre-existing event, occurring after first dose of study treatment.
Additional LNG/EE PK parameters in plasma | Up to Day 21
  Additional LNG/EE PK parameters in plasma.
Povorcitinib concentration in plasma | Up to Day 21
  Povorcitinib concentration in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Celerion Clinical Research Unit, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No